CLINICAL TRIAL: NCT03775109
Title: IL-1 Signal Inhibition in Alcoholic Hepatitis (ISAIAH)
Brief Title: IL-1 Signal Inhibition in Alcoholic Hepatitis
Acronym: ISAIAH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17SM4152; 231612 (Other: IRAS)
Record Dates: First submitted 2018-12-10; First posted 2018-12-13 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Alcoholic Hepatitis
Keywords: Canakinumab; Alcoholic Hepatitis; Alcohol Use Disorder; Interleukin; Treatment; Ilaris; Liver disease
MeSH Terms: conditions — Hepatitis, Alcoholic; Alcoholism; Liver Diseases | interventions — canakinumab; Solutions; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Canakinumab 150mg/ml solution for injection (Active Comparator): 150mg/ml solution for injection
  Interventions: Drug: Canakinumab 150mg/ml solution for injection
- Dextrose (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canakinumab 150mg/ml solution for injection — Canakinumab 150mg/ml solution for injection
  Arms: Canakinumab 150mg/ml solution for injection
Drug: Placebo — 100ml 5% Dextrose
  Arms: Dextrose

SUMMARY:
Alcoholic hepatitis (AH) is a florid presentation of alcoholic liver disease characterized by liver failure in the context of recent and heavy alcohol consumption. The condition carries a high fatality risk; patients with severe AH have a 30% mortality rate at 90 days after presentation.

Currently there is no effective treatment for severe alcoholic hepatitis. Based on the current understanding of the disease pathogenesis IL-1 (interleukin) is a key mediator of hepatic inflammation responsible for metabolic disturbances, fibrogenesis stellate cell activation and consequently portal hypertension.

Canakinumab is a licensed monoclonal antibody inhibitor of IL-1 and may consequently reverse the adverse effects of the cytokine in patients with this disorder. Therefore, the main objective of the ISAIAH trial is to explore the potential benefits of the IL-1β antibody, Canakinumab (solution for injection), in the treatment of alcoholic hepatitis.

ISAIAH is a multicentre, double blind, randomized (1:1), placebo controlled trial. The trial will follow patients up for 90 days and will be conducted in centres across the United Kingdom. Twenty-six patients will be recruited to each arm of the trial: total 52 patients.

DETAILED DESCRIPTION:
The main objective of the ISAIAH trial is to explore the potential benefits of the IL-1β antibody, Canakinumab (solution for injection), in the treatment of alcoholic hepatitis.

ISAIAH is a multicentre, double blind, randomized (1:1), placebo controlled trial. The trial will follow patients up for 90 days and will be conducted in centres across the United Kingdom. Twenty-six patients will be recruited to each arm of the trial: total 52 patients.

The trial will be conducted in patients with severe alcoholic hepatitis (mDF* ≥ 32 and MELD ≤27) with treatment initiated during an index hospital admission with the condition.

The primary endpoint of the trial is histological improvement of alcoholic hepatitis on liver biopsy after 28 days of treatment compared to baseline. Histological improvement is defined as a reduction in lobular inflammation (regardless of cell type).

Patients meeting the eligibility criteria will be randomized and treated. A single dose of 3 mg/kg Canakinumab or identical placebo will be administered intravenously at baseline (Day 1). Canakinumab will be made up by dilution in 100 ml 5% Dextrose by an unblinded research personnel at each site.

Patients with AST >2 x ULN on Day 28 will receive a second dose of 3 mg/kg study drug administered i.v. on Day 28. Patients who received placebo on baseline will receive placebo. Patients who received canakinumab on baseline will receive canakinumab.

Total follow up time for each patient is 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years or older at screening
* Clinical diagnosis of alcoholic hepatitis at screening:

  * Serum bilirubin > 80μmol/L
  * History of excess alcohol (> 80g/day male, > 60g/day female) to within 6 weeks before screening visit
  * Less than 4 weeks since admission to hospital at baseline visit
* mDF* ≥ 32 and MELD ≤ 27 at baseline visit
* Informed consent
* Women of child-bearing potential have to use an effective contraception method (as specified in section 9.6).

Exclusion Criteria:

* Alcohol abstinence of >6 weeks prior to randomization/baseline visit
* Duration of clinically apparent jaundice > 3 months before baseline visit
* Other causes of liver disease including:

  * Evidence of chronic viral hepatitis (Hepatitis B or C)
  * Biliary obstruction
  * Hepatocellular carcinoma
* Evidence of current malignancy (except non-melanotic skin cancer)
* Previous entry into the study, or use of either prednisolone or any systemic steroids (equivalent to a dose of systemic prednisolone >20mg) within 6 weeks of screening.
* AST >500 U/L or ALT >300 U/L (not compatible with alcoholic hepatitis)
* Patients with a serum creatinine >220 μmol/L (2.5 mg / dL) or requiring renal support (see below)
* Patients dependent upon inotropic support (adrenaline or noradrenaline). Terlipressin is allowed
* Variceal haemorrhage on this admission
* Untreated sepsis (see below)
* Patients with known hypersensitivity or contraindications to Canakinumab
* Patients with cerebral haemorrhage, extensive retinal haemorrhage, acute myocardial infarction (within the last 6 weeks) or severe cardiac arrhythmias (not including atrial fibrillation)
* Pregnant or lactating women
* Patients treated with other IL-1 inhibitors and biologics or any other immunosuppressants within 3 months of study participation.
* Known infection with HIV at screening or randomization
* History or evidence of tuberculosis (TB) (active or latent) infection
* Active ongoing inflammatory diseases other than AAH that might confound the evaluation of the benefit of canakinumab therapy
* Underlying metabolic, hematologic, renal, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal conditions, including neutropenia (ANC <1.5) and leukopenia, which in the opinion of the investigator immune-compromises the subject and/or places the subject at unacceptable risk for participation in an immunomodulatory therapy.
* Significant medical problems or diseases, including but not limited to the following: uncontrolled hypertension (≥160/95 mmHg), congestive heart failure [New York Heart Association status of class III or IV], uncontrolled diabetes
* Vaccination with a live vaccine within 3 month before baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Thursz, Study Director — Imperial College London
Locations (16):
- United Kingdom (16):
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Glasgow Royal Infirmary, Greater Glasgow & Clyde, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Aintree University Hospital, Liverpool
  - Royal Liverpool and Broadgreen University Hospitals NHS Trust, Liverpool
  - Imperial College Healthcare NHS Foundation Trust, London
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Royal Free London NHS Foundation Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham
  - John Radcliffe Hospital, Oxford University NHS Foundation Trust, Oxford
  - Plymouth Hospitals NHS Trust, Plymouth
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vergis N, Patel V, Bogdanowicz K, Czyzewska-Khan J, Fiorentino F, Day E, Cross M, Foster N, Lord E, Goldin R, Forrest E, Thursz M. IL-1 Signal Inhibition In Alcoholic Hepatitis (ISAIAH): a study protocol for a multicentre, randomised, placebo-controlled trial to explore the potential benefits of canakinumab in the treatment of alcoholic hepatitis. Trials. 2021 Nov 11;22(1):792. doi: 10.1186/s13063-021-05719-2. PMID 34763711
- [Derived] Vergis N, Patel V, Bogdanowicz K, Czyzewska-Khan J, Keshinro R, Fiorentino F, Day E, Middleton P, Atkinson S, Tranah T, Cross M, Babalis D, Foster N, Lord E, Quaglia A, Lloyd J, Goldin R, Rosenberg W, Parker R, Richardson P, Masson S, Whitehouse G, Sieberhagan C, Patch D, Naoumov N, Dhanda A, Forrest E, Thursz M. IL-1 Signal Inhibition in Alcohol-Related Hepatitis: A Randomized, Double-Blind, Placebo-Controlled Trial of Canakinumab. Clin Gastroenterol Hepatol. 2025 Apr;23(5):797-807.e5. doi: 10.1016/j.cgh.2024.07.025. Epub 2024 Aug 23. PMID 39181422

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 15 sites between February 2019 and October 2020. The first participant was enrolled on 12th February 2019 and the last participant was enrolled on 19th October 2020.
Pre-assignment Details: Of 76 screened participants, 55 met the inclusion criteria and were randomised to treatment.
Groups:
- Canakinumab: A single dose of 3 mg/kg canakinumab administered intravenously at baseline. Canakinumab made up by dilution in 100ml 5% dextrose solution.
  Patients with AST > 2 x ULN on day 28 receive a second dose of 3mg/kg canakinumab administered the same way.
- Placebo: A single injection of 100ml 5% Dextrose solution at baseline.
  Patients with AST > 2 x ULN on day 28 receive a second injection of the same solution.
Period: Overall Study
Arm/Group | Canakinumab | Placebo
Started | 28 | 27
Received First Dose | 27 | 27
Completed | 23 | 23
Not Completed | 5 | 4
Not completed — Adverse Event | 1 | 0
Not completed — COVID-19 outbreak | 2 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canakinumab | Placebo | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (9.1) | 46 (7.8) | 49 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 17 | 13 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 21 | 22 | 43
  Ethnicity: Mixed | 0 | 0 | 0
  Ethnicity: Asian | 4 | 3 | 7
  Ethnicity: Black | 2 | 1 | 3
  Ethnicity: Other | 1 | 1 | 2
Source of patient referral [Count of Participants; unit: Participants]
  GP | 0 | 1 | 1
  A&E | 11 | 15 | 26
  Other hospital | 14 | 11 | 25
  Other | 3 | 0 | 3
Height [Mean (Standard Deviation); unit: cm] | 172 (10.8) | 171 (11.4) | 172 (11.0)
Weight [Mean (Standard Deviation); unit: kg] | 89 (22.2) | 87 (26) | 88 (24.1)
Temperature [Mean (Standard Deviation); unit: Degrees Celsius] | 36.7 (0.25) | 36.7 (0.28) | 36.7 (0.26)
Pulse [Mean (Standard Deviation); unit: BPM] | 81 (13.1) | 85 (11.7) | 83 (12.5)
Systolic BP [Mean (Standard Deviation); unit: mmHg] | 114 (13.4) | 109 (9.9) | 111 (11.9)
Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 68.0 (10.4) | 67 (8.5) | 67 (9.4)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.8 (6.2) | 29.1 (7.1) | 29.5 (6.6)
Physical examination performed [Count of Participants; unit: Participants]
  Yes - abnormalities | 17 | 16 | 33
  Yes - no abnormalities | 6 | 7 | 13
  No | 5 | 4 | 9
WHO Performance Status [Count of Participants; unit: Participants]
  0 - Asymptomatic | 1 | 4 | 5
  1 - Symptomatic but completely ambulatory | 5 | 6 | 11
  2 - Symptomatic < 50% in bed | 7 | 8 | 15
  3 - Symptomatic > 50% in bed | 13 | 9 | 22
  4 - Bedbound | 2 | 0 | 2
Diabetic [Count of Participants; unit: Participants] | 2 | 4 | 6
Previous diagnosis of liver cirrhosis [Count of Participants; unit: Participants]
  Yes - Biopsy | 0 | 1 | 1
  Yes - Clinical | 8 | 6 | 14
  No | 20 | 20 | 40
Previous admission for alcoholic hepatitis [Count of Participants; unit: Participants] | 9 | 4 | 13
Chronic heart disease [Count of Participants; unit: Participants] | 2 | 0 | 2
Chronic lung disease [Count of Participants; unit: Participants] | 0 | 0 | 0
Chronic kidney disease [Count of Participants; unit: Participants] | 1 | 0 | 1
Surgical and medical procedures before entering the study [Count of Participants; unit: Participants] | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Presenting Histological Improvement of Alcoholic Hepatitis on Liver Biopsy After 28 Days of Treatment Compared to Baseline.
Description: Histological improvement is defined as a reduction in lobular inflammation (regardless of cell type).
Time Frame: Baseline and 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 24 | 24
Participants | 14 | 10
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; It is estimated that improvement of histological alcoholic steatohepatitis will occur in 40% of patients treated with placebo and 80% of patients treated with Canakinumab. A trial with 80% power to detect a difference at the P < 0.05 threshold would require 23 patients in each arm, 46 in total. Assuming a drop-out rate of 10%, we will recruit 52 patients in total (26 patients per group); Test type: Superiority; p = 0.248, Chi-squared — The threshold for statistical significance was p = 0.05; Mean Difference (Net) = 16.7, 95% CI 2-sided [-11.2 to 44.5] — Difference = Canakinumab - Placebo

2. Secondary Outcome: Difference in Proportions of Participants With Improvement of Polymorphonuclear Cell Infiltrate From Baseline to Day 28.
Description: Improvement will be recorded as a binary Yes/No outcome. The outcome will be analysed as the proportion of patients, within each treatment group, with improvement on each individual component (polymorphonuclear cell infiltrate, ballooned hepatocytes and steatosis).
Time Frame: Baseline and 28 days
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 23 | 23
Proportion of participants | 0.652 [0.458 to 0.847] | 0.609 [0.409 to 0.808]
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; Mean Difference (Net) = 0.043, 95% CI 2-sided [-0.235 to 0.322] — Difference = Canakinumab - Placebo

3. Secondary Outcome: Number of Patients Presenting Changes in Degree of Fibrosis (AHHS) From Baseline to Day 28
Description: Where presence of bridging fibrosis or Cirrhosis at day 28 is the outcome. Firth logistic regression model was used. An intercept term and treatment indicator are the only predictor variables.
Time Frame: Baseline and 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 23 | 23
Participants | 23 | 22
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; Odds Ratio (OR) = 3.133, 95% CI 2-sided [0.121 to 81.004]

4. Secondary Outcome: Number of Participants Presenting Changes in Steatosis Grade (NAS) From Baseline to Day 28
Description: Number of patients in whom the histological degree of liver steatosis improved between baseline and day 28. Steatosis is assessed using an ordinal scale (1,2,3,4). There are four categories of steatosis grade: (1) <5%, (2) 5% to 33%, (3) >33% to 66%, and (4) >66% Ordinal logistic regression was used for statistical analysis
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 23 | 23
Participants | 15 | 18
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; Odds Ratio (OR) = 1.887, 95% CI 2-sided [0.357 to 9.965]

5. Secondary Outcome: Number of Participants Presenting Changes in Hepatic Venous Pressure Gradient (HVPG) Between Baseline and Day 28
Description: This outcome measure was included in the protocol as a secondary objective. However, no data was generated as HVPG is difficult to obtain and the outcome measure was therefore abandoned
Time Frame: 28 days
Population: No data collected There was no measurement taken
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants Presenting Changes in Serum CK18-M30/M65 From Baseline to Day 7, 14, 21, 28, 42 and 90
Description: Samples were not available. It was reported as a SAP deviation in the final statistical report.
Time Frame: Baseline and 7, 14, 21, 28, 42, 90 days
Population: No data collected Data was not available as samples were not available.
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Serum Bilirubin Concentration From Baseline to Day 28
Time Frame: 28 days
Population: Bilirubin levels at day 28 only.
Measure: Mean (Standard Deviation); unit: micromole/litre
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 25 | 24
micromole/litre | 126 (63.1) | 102 (41.5)
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; p = 0.270, ANCOVA; Change in log-transformed serum bilirubin from baseline to day 28. 49 participants were included in this analysis

8. Secondary Outcome: Change in MELD (Model For End-Stage Liver Disease) Score at From Baseline to Day 28
Description: MELD score is based on the following formula: MELD Score = (9.57 * ln(Creatinine)) + (3.78 * ln(Bilirubin)) + (11.2 * ln(INR)) + 6.43. Higher score is a worse outcome. Minimum value is around 9 and maximum value is around 40.
Time Frame: Day 0 to day 28
Population: Patients with available day 28 MELD score only.
Measure: Mean (Standard Deviation); unit: MELD difference (Units on a scale)
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 25 | 24
MELD difference (Units on a scale) | -4.57 (3.8) | -5.87 (2.9)
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; p = 0.03490, ANCOVA; ANCOVA model: MELD score at Day 28 = intercept + treatment group indicator + baseline MELD score. 49 patients have data at Day 28 and baseline

9. Secondary Outcome: Change in Glasgow Alcoholic Hepatitis Score (GAHS) From Day 28
Description: Predicts mortality in patients with alcoholic hepatitis by laboratory results and age. GAHS score is calculated after Forrest et al., 2007 where a score of 5 to 12 is assigned based on age, WCC, Urea, PT ratio or INR and bilirubin. Higher score means a worse outcome and a score greater than or equal to 9 is associated with a poor prognosis.
  Outcome measure is the score at day 28 - score at day 0
Time Frame: Day 0 to day 28
Population: Patients on whom the Glasgow Alcoholic Hepatitis Score was available at day 28
Measure: Number; unit: score on a scale
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 24 | 24
score on a scale | 1.67 | 1.71
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; Odds Ratio (OR) = 5.088, 95% CI 2-sided [1.558 to 16.624] — Ordinal logistic regression (proportional odds) model. GAHS at day 28 = intercept + treatment group indicator + baseline GAHS measurement. 48 participants have GAHS data at baseline and day 28

10. Secondary Outcome: Change in Maddrey's Discriminant Function (mDF) Score From Baseline to Day 28
Description: mDF is calculated using the following formula: mDF = 4.6 x (Prothrombin time - control time) + Serum Bilirubin (μmol/l) / 17. A higher score is associated with poorer prognosis. A value more than 32 implies poor outcome.
Time Frame: 28 days
Population: Day 28 results.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 25 | 24
score on a scale | 36 (17.7) | 29 (11.4)
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Natural log transformation used for both baseline and day 28 measurements. 49 participants have mDF measurements at baseline and day 28; Test type: Superiority; p = 0.343, ANCOVA; ANCOVA model: mDF score at day 28 = intercept + treatment group indicator + baseline mDF score

11. Secondary Outcome: Lille Score at Day 7
Description: Lille score is calculated as Exp(-R)/[1+exp(-R)] where R = [3.19 - (0.101*age in years)] + (1.47*albumin at baseline in g/dL) + [0.28215* (bilirubin at baseline - bilirubin at Day 8 in mg/dL)] - [0.206 * (if creatinine>=1.3 mg/dL at baseline)] - [0.11115*bilirubin baseline in mg/dL] - (0.0096*Prothrombin Time in seconds at baseline).
  The Lille Model predicts mortality rates within 6 months. Scores >0.45 predict a 6-month survival of 25%. Scores <0.45 predict a 6-month survival of 85%.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 24 | 21
score on a scale | -1.457 (1.085) | -1.540 (0.934)
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; Mean Difference (Net) = 0.083, 95% CI 2-sided [-0.529 to 0.696] — difference = canakinumab - placebo. natural log transformation used

12. Secondary Outcome: Number of Patients With Resolution of Systemic Inflammatory Response Syndrome (SIRS) at Day 28 in Patients With SIRS at Baseline
Description: Recommendations of the American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference; where SIRS represents the presence of 2 or more criteria out of following:
  * Temperature < 36 ºC or > 38 ºC
  * Heart rate > 90 beats/minute
  * Respiratory rate > 20 breaths/minute or venous pCO2 <32 mmHg
  * Leukocyte count > 12,000/mm3 or < 4,000/mm3 or band forms > 10%
Time Frame: 28 days
Population: 6 participants had SIRS at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 2 | 4
Participants | 1 | 3
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact

13. Secondary Outcome: Number of Patients With Incidence of Systemic Inflammatory Response Syndrome (SIRS) at Day 28 in Patients Without SIRS at Baseline
Description: as for outcome 12
Time Frame: 28 days
Population: 43 participants did not have SIRS at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 23 | 20
Participants | 3 | 2
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact

14. Secondary Outcome: Number of Deaths at Day 90
Description: Number of deaths per arm and hazard ratio.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 28 | 27
Participants | 2 | 2
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; Cox Proportional Hazard = 1.046, 95% CI 2-sided [0.147 to 7.424]

15. Secondary Outcome: Number of Patients With Infection Over 90 Days
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 28 | 27
Participants | 6 | 8

16. Secondary Outcome: Number of Patients With Acute Kidney Injury Over 90 Days
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 28 | 27
Participants | 8 | 4

17. Secondary Outcome: Number of Patients With Variceal Haemorrhage Over 90 Days
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 28 | 27
Participants | 1 | 1

18. Secondary Outcome: Number of Participants With Treatment-related Adverse Events
Description: The safety and tolerability of canakinumab will be assessed through the measurement of a number of participants with treatment-related adverse events.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 28 | 27
Participants | 0 | 0

19. Secondary Outcome: Serum and Plasma Biomarkers of Hepatic Function and Inflammation Including Cytokine Profiles Which May Indicate the Degree of Response to IL-1b Inhibition.
Description: Data were not available at time of final analysis.
  The aim is to monitor baseline levels of cytokines linked to inflammasome activation and their changes after active IMP treatment. The proposed method and cytokines is as follows:
  MSD 7-plex kit will be used for the detection of the following cytokines: IL-18, IL-1β*, IL-1ra, IL-6, IL-8, IFNγ** and TNF-α
  ELLA 1-plex will be used for the detection of the following cytokines: IL-18Bpa
Time Frame: 90 days
Population: Data were not available as serum samples required for the cytokine measurements were lost in a freezer failure.
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: CRP Levels at Day 28
Time Frame: 28 days
Population: Number of measurements at day 28
Measure: Median (Inter-Quartile Range); unit: milligrams/litre
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 25 | 24
milligrams/litre | 8 [6.2 to 16] | 10.2 [6.1 to 27]

21. Secondary Outcome: Length of Hospital Stay
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 25 | 26
days | 22 [17 to 34] | 22 [15 to 27]

22. Secondary Outcome: Difference in Proportions of Participants With Improvement of Ballooned Hepatocytes Between Treatment Groups.
Description: Improvement will be recorded as a binary Yes/No outcome. The outcome will be analysed as the proportion of patients, within each treatment group, with 95% confidence intervals.
Time Frame: Day 28
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 23 | 23
Proportion of participants | 0.652 [0.458 to 0.847] | 0.609 [0.409 to 0.808]
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; Mean Difference (Net) = 0.043, 95% CI 2-sided [-0.235 to 0.322] — Difference = Canakinumab - Placebo

23. Secondary Outcome: Difference in Proportions of Improvement of Steatosis Between Treatment Groups at Day 28
Description: as for outcome 22
Time Frame: Day 28
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 23 | 23
Proportion of participants | 0.652 [0.458 to 0.847] | 0.783 [0.614 to 0.951]
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; Mean Difference (Net) = -0.130, 95% CI 2-sided [-0.388 to 0.127] — Difference = Canakinumab - Placebo

24. Secondary Outcome: Number of Patients Presenting Changes in Degree of Neutrophil Infiltration (AHHS) From Baseline to Day 28
Description: Where no/mild polymorphonuclear infiltration at day 28 is the outcome. A logistic regression model was used. An intercept term, baseline measurement and treatment indicator are the only predictor variables.
Time Frame: day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 23 | 23
Participants | 21 | 17
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; Odds Ratio (OR) = 4.012, 95% CI 2-sided [0.693 to 23.219]

25. Secondary Outcome: Number of Patients Presenting Changes in Presence of Megamitochondria (AHHS) From Baseline to Day 28
Description: Where no megamitochondria at day 28 is the outcome. Firth logistic regression model was used. An intercept term, baseline measurement and treatment indicator are the only predictor variables.
Time Frame: day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 23 | 23
Participants | 21 | 19
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; Odds Ratio (OR) = 4.543, 95% CI 2-sided [0.543 to 38.043]

26. Secondary Outcome: Number of Patients Presenting Changes in Type of Bilirubinostasis (AHHS) From Baseline to Day 28
Description: Where there are 3 outcomes: (1) no or hepatocellular only, (2) ductular or canalicular, (3) canalicular or ductular plus hepatocellular. An ordinal logistic regression model was used. An intercept term, baseline measurement and treatment indicator are the only predictor variables.
Time Frame: day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 23 | 23
Participants
  No or hepatocellular only | 14 | 16
  Ductular or canalicular | 3 | 3
  Ductular or canalicular plus Hepatocellular | 6 | 4
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; Odds Ratio (OR) = 1.745, 95% CI 2-sided [0.456 to 6.558]

27. Secondary Outcome: Number of Patients Presenting Changes in Lobular Inflammation (NAS) From Baseline to Day 28
Description: There are four categories: (1) No foci, (2) < 2 foci per 200x field, (3) 2 to 4 foci per 200x field, and (4) > 4 foci per 200x field. Ordinal logistic regression was used.
Time Frame: day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 23 | 23
Participants
  No foci | 1 | 0
  < 2 foci per 200x field | 10 | 14
  2 to 4 foci per 200x field | 11 | 7
  > 4 foci per 200x field | 1 | 2
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; Odds Ratio (OR) = 0.977, 95% CI 2-sided [0.281 to 3.397]

28. Secondary Outcome: Number of Patients Presenting Changes in Hepatocyte Ballooning (NAS) From Baseline to Day 28
Description: There are three categories: (1) none, (2) few balloon cells, and (3) many cells/prominent ballooning. Ordinal logistic regression was used.
Time Frame: day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 23 | 23
Participants
  None | 1 | 3
  Few balloon cells | 15 | 11
  Many cells/prominent ballooning | 7 | 9
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; Odds Ratio (OR) = 0.768, 95% CI 2-sided [0.238 to 2.479]

29. Secondary Outcome: Number of Patients With Sepsis Over 90 Days
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 28 | 27
Participants | 1 | 1

30. Secondary Outcome: Number of Patients With Ascites Over 90 Days
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 28 | 27
Participants | 26 | 21

31. Secondary Outcome: Number of Patients With Encephalopathy Over 90 Days
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 28 | 27
Participants | 9 | 6

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Canakinumab | Placebo
All-Cause Mortality (participants affected / at risk) | 2/28 | 2/27
Serious Adverse Events (participants affected / at risk) | 10/28 | 10/27
Other Adverse Events (participants affected / at risk) | 26/28 | 24/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Canakinumab (N=28) | Placebo (N=27)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Alcoholic liver disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ascites (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 4 (5)
Hepatic encephalopathy (Hepatobiliary disorders) | 2 (2) | 0 (0)
Oesophageal varices haemorrhage (Hepatobiliary disorders) | 1 (2) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Haemoperitoneum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Soft tissue necrosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Canakinumab (N=28) | Placebo (N=27)
General AE (General disorders) | 26 (114) | 24 (102)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT03775109/Prot_SAP_000.pdf